CLINICAL TRIAL: NCT05186246
Title: Effectivity and Safety of Combination of Spent Grain Wax, Argan Oil, Shea Butter and Saccharide Isomerate Post Fractional CO2 Laser
Brief Title: Effectivity and Safety of Combination of Spent Grain Wax, Argan Oil, Shea Butter and Saccharide Isomerate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr.dr.Irma Bernadette, SpKK (K) (Other)
Responsible Party: Sponsor-Investigator, Dr.dr.Irma Bernadette, SpKK (K), Dr. dr. Irma Bernadette S. Sitohang, SpKK(K) - Head of Cosmetic Dermatology Division of Dermatology and Venereology Department of Faculty of Medicine Universitas Indonesia / Cipto Mangunkusumo Hospital, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EffectivityCombiSpentGrain
Record Dates: First submitted 2021-12-13; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Acne Vulgaris
Keywords: laser; cream; fractional co2 laser; spent wax
MeSH Terms: conditions — Acne Vulgaris | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Combination Cream Group (Experimental): Subjects were randomized to have combination cream to be applied on one side of the face twice daily post fractional CO2 laser. The subjects were evaluated on day 3 and day 7 post fractional CO2 laser. Combination cream consisted of Spent Grain Wax, Argan Oil, Shea Butter and Saccharide Isomerate cream
  Interventions: Drug: Combination cream
- Placebo comparator (Placebo Comparator): Subjects were randomized to have placebo cream to be applied on the other side of the face twice daily post fractional CO2 laser. Placebo cream were packaged in identical-looking containers with combination cream. The subjects were evaluated on day 3 and day 7 post fractional CO2 laser.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Combination cream — Spent Grain Wax, Argan Oil, Shea Butter and Saccharide Isomerate Cream combination (10 gram), were applied on one side of the face twice daily by participants.
  Arms: Experimental Combination Cream Group
Drug: Placebo cream — Cream that is identical looking were given to subjects to be applied on the other side of the face twice daily
  Arms: Placebo comparator

SUMMARY:
The clinical study will compare the efficacy and safety of Combination of Spent Grain Wax, Argan Oil, Shea Butter and Saccharide Isomerate cream post fractional CO2 laser. Combination of Spent Grain Wax, Argan Oil, and Shea Butter was formulated to reduce skin irritation and allergy symptoms such as dryness, itch and rash. The combination cream applied on one side of the face while placebo will be applied on the other side of the face in 18-60 years old female post fractional CO2 laser.

DETAILED DESCRIPTION:
This study is an experimental study with a randomized controlled trial (RCT) design on patients who met the inclusion criteria. All participants will receive pretreatment in the form of 0.05% tretinoin cream for two weeks, then all participants will undergo fractional CO2 laser treatment. Post laser treatment, the participants will be given cream A and B, which already randomized to be applied on to the face. All participants will be evaluated in day 3 and day 7 post fractional CO2 laser. The results of therapy will mainly be assessed based on the Dermoscopic Photoaging Scale (DPAS), as well as visual analog scale (VAS) for subjective symptoms and Clinician Erythema Assessment Scale (CEA) for erythema and Skin Capacitance measured with TEWAmeter.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-60 years old with an understanding of all the information given by written consent form
* Had undergone priming with tretinoin cream 0,05% for 2 weeks pre fractional CO2 laser treatment

Exclusion Criteria:

* Personal or family history of skin cancer, especially melanoma
* Consumption of systemic retinoic acid within 3 month of enrollment
* Use of any topical skin brightening or whitening preparations within 1 month of enrollment
* Pigmentary disorders or any dermatoses, which may affect the measurement within the study areas
* A pregnant or breastfeeding mother
* History of hormonal or endocrine diseases or taking medication for hormonal or endocrine diseases
* Inability to comply research protocols

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of Eryhtema Score | baseline; 3 days post fractional CO2 laser; and 7 days post fractional CO2 laser
  Based on Clinical Erythema Assessment Scale. Scale range is 0-4, 0 indicates no erythema and 4 indicates severe erythema
Change of Photoaging Skin Condition | baseline; 3 days post fractional CO2 laser; and 7 days post fractional CO2 laser
  This DPAS assessment is based on yes or no rules on 11 criteria in four facial regions, namely left malar, right malar, forehead, and chin. The criteria were yellowish discoloration, white line, lentigo, hypo- and hyper-pigmented macules, telangiectasia, yellow papules, actinic keratosis, senile comedones, deep wrinkle, superficial wrinkle, and criss-cross wrinkle. Score range is 0-44 points.
Change of Subjective Pain Evaluation | baseline; 3 days post fractional CO2 laser; and 7 days post fractional CO2 laser
  Assessed using Visual Analog Scale (VAS). Scale range is 0-10, 0 indicates no pain and 10 indicates severe pain
Change of Skin Capacitance | baseline; 3 days post fractional CO2 laser; and 7 days post fractional CO2 laser
  Assessed using TEWAmeter to see changes in Skin Capacitance
Change of Skin Conditions of patients assessed by Janus Facial Analysis System | baseline; 3 days post fractional CO2 laser; and 7 days post fractional CO2 laser
  Assessed using Janus Facial Analysis System® Skin will be assessed using Janus with three different wavelength of light which are normal, polarized and UV light. The skin will be analyzed for pores, wrinkles, sebum and skin tone

CONTACTS AND LOCATIONS:
Overall Officials: Irma BS Sitohang, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Rumah Sakit Angkatan Darat Gatot Soebroto, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No